CLINICAL TRIAL: NCT05131646
Title: Extension Study to Evaluate the Long-term Outcomes of Subjects Following CLS-AX Administration for Age-related Macular Degeneration in the CLS-AX CLS1002-101 Study
Brief Title: Extension Study to Evaluate the Long-term Outcomes of Subjects in the CLS-AX CLS1002-101 Study
Status: Completed | Type: Observational
Sponsor: Clearside Biomedical, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CLS1002-102
Record Dates: First submitted 2021-10-26; First posted 2021-11-23 (Actual); Results first posted 2024-03-04 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2023-02

CONDITIONS: Neovascular Age-related Macular Degeneration
Keywords: AMD; Wet-AMD; suprachoroidal; tyrosine kinase inhibitor; nAMD; SCS

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cohort 2 (Low-mid Dose) Extension: Subjects who were administered by suprachoroidal injection 0.10 mg CLS-AX in cohort 2 of the parent study, CLS1002-101, will be followed for an additional 12 weeks following exit from the Parent study. No intervention will be administered in this extension study.
  Interventions: Drug: CLS-AX
- Cohort 3 (High-mid Dose) Extension: Subjects who were administered by suprachoroidal injection 0.50 mg CLS-AX in cohort 3 of the parent study, CLS1002-101, will be followed for an additional 12 weeks following exit from the Parent study. No intervention will be administered in this extension study.
  Interventions: Drug: CLS-AX
- Cohort 4 (High Dose) Extension: Subjects who were administered by suprachoroidal injection 1.0 mg CLS-AX in cohort 4 of the parent study, CLS1002-101, will be followed for an additional 12 weeks following exit from the Parent study. No intervention will be administered in this extension study.
  Interventions: Drug: CLS-AX

INTERVENTIONS:
Drug: CLS-AX — injectable suspension of small molecule tyrosine kinase inhibitor (TKI) administered in the Parent study CLS1002-101
  Other Names: axitinib injectable suspension

SUMMARY:
This is an open-label, non-interventional extension study of up to 12 weeks in duration in subjects completing Cohorts 2, 3, and 4 of the Parent study, CLS1002-101.

DETAILED DESCRIPTION:
This is an open-label, non-interventional extension study of up to 12 weeks in duration in subjects completing Cohorts 2. 3 and 4 of the Parent study, CLS1002-101. The Parent study is a 12-week, Phase 1/2a, multicenter study designed to assess the safety and tolerability of a single dose of CLS-AX administered suprachoroidally in subjects with neovascular age-related macular degeneration (nAMD) who show stable visual acuity following 3 or more injections with an intravitreal (IVT) anti-VEGF therapy in the preceding 5 months.

Summary analyses will include 12-weeks data from the Parent study, CLS1002-101, and 12-weeks data from this extension study, CLS1002-102, for a total of 24 weeks follow-up, for all participants enrolled into the extension study.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in and completed the Parent study, CLS1002-101, as part of Cohort 2 or Cohort 3 or Cohort 4.

Exclusion Criteria:

* Received prohibited medication in the Parent study, CLS1002-101.
* Enrolled in the Parent study CLS1002-101 as part of Cohort 1.
* Females of childbearing potential who are pregnant and or lactating.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants who completed cohort 2 or 3 or 4 of CLS1002-101
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2021-10-08 (Actual); Primary Completion 2023-01-05 (Actual); Study Completion 2023-01-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Coultas, PhD, Study Director — Clearside Biomedical, Inc.
Locations (7):
- United States (7):
  - Retinal Consultants of Arizona, Phoenix, Arizona
  - Northern California Retina Vitreous Associates Medical Group, LLC, Mountain View, California
  - Retina Consultants Medical Group, Inc, Sacramento, California
  - Southeast Retina Center, Augusta, Georgia
  - Cumberland Valley Retina Consultants, Hagerstown, Maryland
  - Retina Consultants of Texas, Bellaire, Texas
  - Retina Consultants of Texas, The Woodlands, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cohort 2 (Low-mid Dose) Extension | Cohort 3 (High-mid Dose) Extension | Cohort 4 (High Dose) Extension
Started | 3 | 7 | 5
Safety Population | 3 | 7 | 5
Completed | 2 | 7 | 5
Not Completed | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 2 (Low-mid Dose) Extension | Cohort 3 (High-mid Dose) Extension | Cohort 4 (High Dose) Extension | Total
Number analyzed (Participants) | 3 | 7 | 5 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 78.7 (9.02) | 87.9 (4.98) | 79.6 (3.97) | 83.3 (6.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 4 | 11
  Male | 1 | 2 | 1 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 7 | 5 | 15
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 3 | 7 | 5 | 15
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 7 | 5 | 15
Duration of nAMD Diagnosis in the Study Eye [Mean (Standard Deviation); unit: months] | 56.63 (23.759) | 67.29 (44.329) | 36.42 (38.955) | 54.87 (39.442)
Total Number of Prior nAMD Treatments in the Study Eye [Count of Participants; unit: Participants]
  0-2 Injections | 0 | 0 | 0 | 0
  3-6 Injections | 0 | 2 | 1 | 3
  7-12 Injections | 1 | 0 | 1 | 2
  13-18 Injections | 0 | 1 | 0 | 1
  >18 Injections | 2 | 4 | 3 | 9
Pre Injection Intraocular Pressure in the Study Eye at Baseline [Mean (Standard Deviation); unit: mmHg] — Intraocular pressure (IOP) is a diagnostic measurement of the fluid pressure, measured in millimeters of mercury, inside the eye. IOP was measured using Goldmann applanation tonometry or by use of a Tonopen tonometer. Normal eye pressure is usually considered to be between 10 and 20 mmHg (AAO.org). Untreated elevated eye pressure is a risk factor for glaucoma.
  mmHg | 14.3 (1.53) | 13.9 (2.34) | 13.8 (3.56) | 13.9 (2.52)
Best Corrected Visual Acuity in the Study Eye at Baseline [Mean (Standard Deviation); unit: letters] — Best corrected visual acuity (BCVA) at a starting distance of 4 meters. The BCVA letter score ranges from 0 to 100 (best score attainable), with a higher score indicating better visual acuity.
  letters | 61.0 (8.19) | 59.0 (14.71) | 71.2 (2.17) | 63.5 (11.67)
Central Subfield Thickness in the Study Eye at Baseline [Mean (Standard Deviation); unit: microns] — Central subfield thickness (CST) is a diagnostic measurement used in identifying the presence of edema in the circular area 1 mm in diameter centered around the fovea. CST was measured using spectral domain optical coherence tomography (SD-OCT). A central reading center graded the SD-OCT digital images. Only images that were gradable by the central reading center were included in the analysis.
  microns | 214.0 (13.53) | 201.9 (24.38) | 214.8 (13.74) | 208.6 (19.43)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: The number of participants with treatment-emergent adverse events (TEAEs) reported between the administration of CLS-AX and study exit.
Time Frame: Day 1 to Week 24
Population: Defined as all enrolled participants who were administered CLS-AX in the Parent study, who have provided informed consent for participating in the Extension study, and from whom at least one safety measurement was obtained after the participant provided informed consent.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2 (Low-mid Dose) Extension | Cohort 3 (High-mid Dose) Extension | Cohort 4 (High Dose) Extension
Number analyzed (Participants) | 3 | 7 | 5
Participants | 3 | 2 | 1

2. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: The number of participants with serious adverse events (SAEs) reported between the administration of CLS-AX and study exit.
Time Frame: Day 1 to Week 24
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2 (Low-mid Dose) Extension | Cohort 3 (High-mid Dose) Extension | Cohort 4 (High Dose) Extension
Number analyzed (Participants) | 3 | 7 | 5
Participants | 0 | 0 | 0

3. Secondary Outcome: Mean Change From Baseline in Central Subfield Thickness (CST) in the Study Eye
Description: Central subfield thickness (CST) is a diagnostic measurement used in identifying the presence of edema in the circular area 1 mm in diameter centered around the fovea. CST was measured using spectral domain optical coherence tomography (SD-OCT). A central reading center graded the SD-OCT digital images. A negative change from baseline value represents a reduction in macular edema. Only images that were gradable by the central reading center were included in the analysis.
Time Frame: Weeks 4, 8, 12, 16, 20 and 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: microns
Arm/Group | Cohort 2 (Low-mid Dose) Extension | Cohort 3 (High-mid Dose) Extension | Cohort 4 (High Dose) Extension
Number analyzed (Participants) | 3 | 7 | 5
microns
  Week 4: number analyzed (Participants) | 3 | 6 | 5
  Week 4 | 14.7 (14.47) | 23.5 (23.82) | 20.2 (26.64)
  Week 8: number analyzed (Participants) | 3 | 6 | 5
  Week 8 | 5.7 (30.37) | 28.2 (21.48) | 13.6 (18.08)
  Week 12 | 53.3 (83.34) | 36.6 (34.02) | 19.4 (16.10)
  Week 16: number analyzed (Participants) | 2 | 7 | 5
  Week 16 | 18.0 (19.80) | 5.1 (28.26) | 13.4 (15.49)
  Week 20: number analyzed (Participants) | 1 | 7 | 5
  Week 20 | 67.0 | 20.0 (21.84) | 26.2 (49.55)
  Week 24: number analyzed (Participants) | 1 | 7 | 5
  Week 24 | 6.0 | 20.4 (33.10) | 26.4 (65.26)

4. Secondary Outcome: Mean Change From Baseline in Best Corrected Visual Acuity (BCVA) Letter Score in the Study Eye
Description: BCVA measured on the Early Treatment Diabetic Retinopathy Study (ETDRS) chart at a starting test distance of 4 meters. The BCVA letter score ranges from 0 to 100 (best score attainable), and a gain in BCVA letter score from baseline indicates an improvement in visual acuity.
Time Frame: Weeks 4, 8, 12, 16, 20 and 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | Cohort 2 (Low-mid Dose) Extension | Cohort 3 (High-mid Dose) Extension | Cohort 4 (High Dose) Extension
Number analyzed (Participants) | 3 | 7 | 5
letters
  Week 4: number analyzed (Participants) | 3 | 6 | 5
  Week 4 | 0.7 (2.08) | 1.0 (2.19) | 0.8 (2.49)
  Week 8: number analyzed (Participants) | 3 | 6 | 5
  Week 8 | -2.3 (2.08) | 2.5 (3.08) | 1.8 (2.86)
  Week 12 | -5.0 (10.82) | -0.9 (2.85) | 0.0 (3.16)
  Week 16: number analyzed (Participants) | 2 | 7 | 5
  Week 16 | -2.0 (0.00) | 1.9 (3.02) | 1.0 (4.85)
  Week 20: number analyzed (Participants) | 2 | 7 | 5
  Week 20 | 0.0 (1.41) | 0.0 (2.65) | 1.0 (6.20)
  Week 24: number analyzed (Participants) | 2 | 7 | 5
  Week 24 | -35.0 (46.67) | -1.9 (5.05) | 0.4 (6.62)

5. Secondary Outcome: Number of Participants Receiving Additional Intravitreal (IVT) Aflibercept Injections
Description: Number of participants receiving additional intravitreal aflibercept injections during the course of the study for nAMD.
Time Frame: Day 1 to Week 24
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2 (Low-mid Dose) Extension | Cohort 3 (High-mid Dose) Extension | Cohort 4 (High Dose) Extension
Number analyzed (Participants) | 3 | 7 | 5
Participants
  Week 4: number analyzed (Participants) | 3 | 6 | 5
  Week 4 | 1 | 0 | 1
  Week 8: number analyzed (Participants) | 3 | 6 | 5
  Week 8 | 1 | 0 | 0
  Week 12 | 1 | 1 | 1
  Week 16: number analyzed (Participants) | 2 | 7 | 5
  Week 16 | 0 | 0 | 0
  Week 20: number analyzed (Participants) | 2 | 7 | 5
  Week 20 | 1 | 0 | 2
  Week 24: number analyzed (Participants) | 2 | 7 | 5
  Week 24 | 0 | 2 | 1
  Day 1 to Week 24 | 3 | 2 | 3

6. Other Pre Specified Outcome: Number of Participants Qualifying to Receive Additional Intravitreal (IVT) Aflibercept Injections
Description: Number of participants qualifying to receive additional intravitreal aflibercept injections during the course of the study. Criteria included 1) loss of 10 or more letters in BCVA compared to the best prior study-assessed BCVA in the study eye that was attributed to intra- or sub-retinal fluid, 2) increase in central subfield thickness >75 microns from Baseline in the study eye, or 3) presence of vision-threatening hemorrhage due to AMD in the study eye.
Time Frame: Day 1 to Week 24
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2 (Low-mid Dose) Extension | Cohort 3 (High-mid Dose) Extension | Cohort 4 (High Dose) Extension
Number analyzed (Participants) | 3 | 7 | 5
Participants
  Week 4: number analyzed (Participants) | 3 | 6 | 5
  Week 4 | 1 | 0 | 1
  Week 8: number analyzed (Participants) | 3 | 6 | 5
  Week 8 | 1 | 0 | 0
  Week 12 | 1 | 1 | 1
  Week 16: number analyzed (Participants) | 2 | 7 | 5
  Week 16 | 0 | 0 | 0
  Week 20: number analyzed (Participants) | 2 | 7 | 5
  Week 20 | 1 | 0 | 2
  Week 24: number analyzed (Participants) | 2 | 7 | 5
  Week 24 | 1 | 2 | 1
  Day 1 to Week 24 | 3 | 2 | 3

7. Other Pre Specified Outcome: Mean Change From Baseline in Pre-Injection Intraocular Pressure (IOP)
Description: Intraocular pressure (IOP) is a diagnostic measurement of the fluid pressure, measured in millimeters of mercury, inside the eye. IOP was measured using Goldmann applanation tonometry or by use of a Tonopen tonometer. Normal eye pressure is usually considered to be between 10 and 20 mmHg (AAO.org). Untreated elevated eye pressure is a risk factor for glaucoma.
Time Frame: Weeks 4, 8, 12, 16, 20 and 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Cohort 2 (Low-mid Dose) Extension | Cohort 3 (High-mid Dose) Extension | Cohort 4 (High Dose) Extension
Number analyzed (Participants) | 3 | 7 | 5
mmHg
  Week 4: number analyzed (Participants) | 3 | 6 | 5
  Week 4 | -0.7 (4.16) | -0.5 (0.84) | 0.2 (5.45)
  Week 8: number analyzed (Participants) | 3 | 6 | 5
  Week 8 | 0.3 (3.79) | 0.2 (1.72) | 1.6 (3.78)
  Week 12 | 0.3 (2.31) | -0.1 (1.68) | 0.2 (3.90)
  Week 16: number analyzed (Participants) | 2 | 7 | 5
  Week 16 | 0.5 (3.54) | 0.4 (1.72) | 1.2 (2.49)
  Week 20: number analyzed (Participants) | 2 | 7 | 5
  Week 20 | 1.0 (0.00) | -0.6 (0.98) | 0.0 (3.54)
  Week 24: number analyzed (Participants) | 2 | 7 | 5
  Week 24 | -1.0 (4.24) | 0.6 (1.99) | 0.4 (3.91)

ADVERSE EVENTS:
Time Frame: Adverse events were collected over 24 weeks following CLS-AX administration.
Arm/Group | Cohort 2 (Low-mid Dose) Extension | Cohort 3 (High-mid Dose) Extension | Cohort 4 (High Dose) Extension
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/7 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/7 | 0/5
Other Adverse Events (participants affected / at risk) | 3/3 | 2/7 | 1/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 2 (Low-mid Dose) Extension (N=3) | Cohort 3 (High-mid Dose) Extension (N=7) | Cohort 4 (High Dose) Extension (N=5)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0) — Study eye
Conjunctival oedema (Eye disorders) | 0 (0) | 1 (1) | 0 (0) — Study eye
Macular degeneration (Eye disorders) | 1 (2) | 0 (0) | 0 (0) — Study eye
Neovascular age-related degeneration (Eye disorders) | 0 (0) | 1 (1) | 0 (0) — Study eye
Retinal haemorrhage (Eye disorders) | 1 (1) | 1 (1) | 0 (0) — Study eye
Subretinal fluid (Eye disorders) | 1 (1) | 0 (0) | 0 (0) — Study eye
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All information concerning CLS1002-102 and the operations of Clearside Biomedical, Inc. are considered CONFIDENTIAL and shall remain the sole property of Clearside Biomedical Inc. The institutions and Investigators participating in this study shall have no right to publish or present the results of this study without the prior written consent of Clearside Biomedical, Inc.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-26): https://cdn.clinicaltrials.gov/large-docs/46/NCT05131646/Prot_SAP_000.pdf